CLINICAL TRIAL: NCT00027573
Title: Adoptive Immunotherapy by Allogeneic Stem Cell Transplantation for Metastatic Renal Cell Carcinoma: A Phase II Study
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-90003; U10CA031946 (NIH); CALGB-90003; CDR0000069044 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma; papillary renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Filgrastim; Cyclophosphamide; fludarabine phosphate; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy + stem cell transplantation (Experimental): Patients receive fludarabine IV over 30 minutes on days -7 to -3 and cyclophosphamide IV over 1-2 hours on days -4 and -3. Allogeneic peripheral blood stem cells are infused on day 0. Patients then receive filgrastim (G-CSF) subcutaneously daily beginning on day 5 and continuing until blood counts recover.
  Patients receive graft-versus-host disease (GVHD) prophylaxis comprising oral tacrolimus twice daily on days -1 to 90 and methotrexate IV on days 1, 3, and 6.
  After day 120, patients with persistent disease and no signs of active GVHD may receive donor lymphocyte infusion (DLI). DLI may be repeated every 8 weeks for a total of 2 infusions.
  Patients are followed every 2 months for 1 year and then every 6 months for 4 years OR every 2 months for 6 months and then every 6 months for 4.5 years if patient receives DLI.
  Interventions: Biological: filgrastim; Biological: therapeutic allogeneic lymphocytes; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: methotrexate
Drug: tacrolimus
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by donor peripheral stem cell transplantation in treating patients who have metastatic or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate and overall and disease-free survival of patients with unresectable or metastatic renal cell cancer treated with fludarabine and cyclophosphamide followed by allogeneic peripheral blood stem cell transplantation.
* Determine the toxicity and treatment-related mortality of this regimen in these patients.
* Determine the percentage of donor chimerism in patients treated with this regimen.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma (RCC)

  * Clear cell or papillary RCC
  * Granular tumors with sarcomatoid features
  * No purely sarcomatoid RCC, chromophobic RCC, or oncocytoma
  * No transitional cell carcinoma of the renal pelvis and collecting systems
* Metastatic or unresectable disease
* At least 1 measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Primary bladder masses
* Progressive disease after interferon alfa and/or interleukin-2 for metastatic RCC OR intolerance to these therapies
* No prior or concurrent CNS metastases

  * Negative MRI of the brain within the past 28 days
* Must have HLA-identical (6/6) sibling donor

PATIENT CHARACTERISTICS:

Age:

* 60 and under

Performance status:

* ECOG 0-1

Life expectancy:

* More than 6 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine clearance at least 40 mL/min

Cardiovascular:

* LVEF at least 45% by MUGA or echocardiogram

Pulmonary:

* DLCO greater than 40% of predicted (corrected for hemoglobin level)
* No symptomatic pulmonary disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No known hypersensitivity to E. coli-derived products
* No uncontrolled diabetes mellitus
* No active serious infection
* No other concurrent malignancy except non-melanoma skin cancer or other malignancy that has less than a 30% risk of relapse after completion of therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent sargramostim (GM-CSF)
* Concurrent epoetin alfa allowed

Chemotherapy:

* No other concurrent chemotherapy

Endocrine therapy:

* At least 28 days since prior hormonal therapy (e.g., megestrol, corticosteroids, or anti-estrogen therapy)
* Concurrent steroids allowed for adrenal failure, graft-versus-host disease, or other nondisease-related conditions (e.g., insulin for diabetes)

Radiotherapy:

* At least 14 days since prior radiotherapy

Surgery:

* At least 14 days since prior surgery

Other:

* At least 28 days since prior systemic therapy for RCC
* Recovered from prior therapy

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2001-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 5 years
Overall survival | Up to 5 years
Disease-free survival | Up to 5 years
Treatment-related mortality | Up to 5 years
Percentage of donor chimerism in patients treated | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian I. Rini, MD, Study Chair — University of California, San Francisco
Locations (6):
- United States (6):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - CCOP - Oklahoma, Tulsa, Oklahoma

REFERENCES:
- [Result] Rini BI, Halabi S, Barrier R, Margolin KA, Avigan D, Logan T, Stadler WM, McCarthy PL, Linker CA, Small EJ; Cancer and Leukemia Group B; Eastern Cooperative Oncology Group; Southwestern Oncology Group. Adoptive immunotherapy by allogeneic stem cell transplantation for metastatic renal cell carcinoma: a CALGB intergroup phase II study. Biol Blood Marrow Transplant. 2006 Jul;12(7):778-85. doi: 10.1016/j.bbmt.2006.03.011. PMID 16785067